CLINICAL TRIAL: NCT03498651
Title: Effectiveness of Interpretation of Training to Reduce Anxiety: Evaluating Technology-based Delivery Models and Methods to Reduce Attrition
Brief Title: Interpretation Training to Reduce Anxiety: Evaluating Technology-based Delivery Models and Methods to Reduce Attrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bethany A. Teachman, Ph.D., Professor, University of Virginia
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0234-00
Record Dates: First submitted 2018-03-31; First posted 2018-04-17 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Anxiety
Keywords: Anxiety; Cognitive bias; Telemedicine
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Participants will be aware whether they are completing the intervention by phone or computer, and will know if they are receiving coaching or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBM-I, low attrition (Experimental): Computer- or phone-based Cognitive Bias Modification - Interpretation training
  Interventions: Behavioral: Cognitive Bias Modification - Interpretation training
- CBM-I, high attrition, coach (Experimental): Computer- or phone-based Cognitive Bias Modification - Interpretation training + Coaching
  Interventions: Behavioral: Cognitive Bias Modification - Interpretation training; Behavioral: Coaching
- CBM-I, high attrition, no coach (Experimental): Computer- or phone-based Cognitive Bias Modification - Interpretation training
  Interventions: Behavioral: Cognitive Bias Modification - Interpretation training
- Psychoeducation (Active Comparator): Online psychoeducation about anxiety
  Interventions: Behavioral: Online psychoeducation about anxiety

INTERVENTIONS:
Behavioral: Cognitive Bias Modification - Interpretation training — Training involves presenting participants with brief scenarios that introduce an ambiguous potential threat. Critically, the ambiguity regarding how the situation is resolved remains until the last word of the scenario, which is presented as a word fragment that the participant must solve, which will typically then assign a benign (rather than threatening) meaning to the scenario.
  Arms: CBM-I, high attrition, coach; CBM-I, high attrition, no coach; CBM-I, low attrition
Behavioral: Coaching — Participants identified as high risk for attrition will receive low-intensity coaching, which includes a mix of brief phone calls, texts, and/or emails with a trained member of the study team to help address challenges with adherence to and application of the training.
  Arms: CBM-I, high attrition, coach
Behavioral: Online psychoeducation about anxiety — Participants will review webpages that describe information about symptoms and causes of anxiety, including the nature of biased thinking in anxiety.
  Arms: Psychoeducation

SUMMARY:
The project aims to compare effectiveness and target engagement of CBM-I delivered via computer vs. mobile phone, and test if adding minimal human contact for participants at risk of dropout improves retention and outcomes.

DETAILED DESCRIPTION:
Approximately 25-30% of the U.S. population will experience anxiety pathology severe enough to qualify for an anxiety disorder diagnosis during their lifetime. Critically, the majority will not receive treatment, creating a serious need to consider alternative approaches to delivering mental health services that can meet needs on a larger scale. Cognitive Bias Modification (CBM) interventions for anxiety hold considerable promise as a way to meet these needs. These programs alter biased ways of thinking, such as selective assignment of threat interpretations, which are known to cause and maintain anxiety. CBM for interpretation bias (CBM-I) has established efficacy when administered via computer in the laboratory, and there is clear evidence for target engagement (i.e., change in interpretations, the identified mechanism). Now, effectiveness needs to be tested in the community, using sufficiently large samples to evaluate key moderators of its effects, including delivery method (computer vs. mobile phone) and the addition of minimal human contact (for those at risk of attrition). Addressing attrition is critical given high rates of drop out for web-based interventions. Via the PI's MindTrails web site (established with the lab's prior NIMH R34MH106770 award), the lab already has the infrastructure to deliver CBM to the public and recruit large anxious samples. Moreover, the PI and Co-I have established infrastructure to do mobile sensing of mood and CBM-I delivery via mobile phones. Thus, the project can respond to NIMH's request for "Effectiveness trials that can contribute to advancing the personalization of mental health care." The current proposal aims to compare effectiveness and target engagement of CBM-I delivered via computer vs. mobile phone, and test if adding minimal human contact for participants at risk of dropout improves retention and outcomes. Study 1 will provide a pilot feasibility and user experience test of the CBM-I program on mobile phones. Study 2 will examine the lab's current online, computer-based CBM-I data to help determine empirical indicators of attrition. Study 3 will provide the primary test of moderators of effectiveness. Namely, in Study 3, high anxious participants will be randomized to one of 2 conditions: 1) CBM-I training delivered by computer or mobile phone (at existing MindTrails site); 2) Alternate intervention group-Psychoeducation only. CBM-I and Psychoeducation conditions include 5 weekly training sessions. Based on theoretically- and empirically-derived predictors of attrition, participants identified as high-risk for dropout in condition 1 will then be randomly assigned to add minimal human contact (using a modified TeleCoach protocol) or no change. Using this adaptive intervention, known as Sequential, Multiple Assignment, Randomized Trial (SMART), the project can test both the effects of CBM-I delivery method and the added value of human contact to improve retention for participants at high-risk for dropping out.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Moderate to extremely severe anxiety range (i.e., 10 or higher) on the Depression, Anxiety, Stress Scales - Short Form: Anxiety Subscale
* Regular access to the Internet via Smartphone or computer

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1748 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Teachman, PhD, Principal Investigator — Univ. of Virginia
Locations (1):
- MindTrails web site: https://mindtrails.virginia.edu/ (thru Univ. of Virginia), Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on the NIMH Data Archive.
Time Frame: Data will be shared within one year of completion of the main trial.
Access Criteria: We will follow the standard access criteria for the NIMH Data Archive.
URL: https://data-archive.nimh.nih.gov/

REFERENCES:
- [Derived] Eberle JW, Daniel KE, Baee S, Silverman AL, Lewis E, Baglione AN, Werntz A, French NJ, Ji JL, Hohensee N, Tong X, Huband JM, Boukhechba M, Funk DH, Barnes LE, Teachman BA. Web-based interpretation bias training to reduce anxiety: A sequential, multiple-assignment randomized trial. J Consult Clin Psychol. 2024 Jun;92(6):367-384. doi: 10.1037/ccp0000896. PMID 39023984

RESULTS

PARTICIPANT FLOW:
Groups:
- Received CBM-I and Not Classified as High/Low Risk for Attrition: This group started treatment (and had been Stage 1 randomized to CBM-I) but did not complete Session 1 of CBM-I training plus assessments, so was not classified as high/low risk for attrition and thus not randomized for Stage 2 of SMART design
- Received CBM-I and Classified Low Attrition; Received CBM-I and Classified High Attrition and no Coach Given: Computer- or phone-based Cognitive Bias Modification - Interpretation training
  Cognitive Bias Modification - Interpretation training: Training involves presenting participants with brief scenarios that introduce an ambiguous potential threat. Critically, the ambiguity regarding how the situation is resolved remains until the last word of the scenario, which is presented as a word fragment that the participant must solve, which will typically then assign a benign (rather than threatening) meaning to the scenario.
- Received CBM-I and Classified High Attrition and Given a Coach: Computer- or phone-based Cognitive Bias Modification - Interpretation training + Coaching
  Cognitive Bias Modification - Interpretation training: Training involves presenting participants with brief scenarios that introduce an ambiguous potential threat. Critically, the ambiguity regarding how the situation is resolved remains until the last word of the scenario, which is presented as a word fragment that the participant must solve, which will typically then assign a benign (rather than threatening) meaning to the scenario.
  Coaching: Participants identified as high risk for attrition will receive low-intensity coaching, which includes a mix of brief phone calls, texts, and/or emails with a trained member of the study team to help address challenges with adherence to and application of the training.
- Psychoeducation, Lacking Classification Measures: This group started treatment (and had been Stage 1 randomized to psychoeducation) but did not complete Session 1 of psychoeducation plus assessments, so is not part of the classification measure completer sample
- Not Randomized to Treatment: Completed consent but didn't complete baseline assessments or reach point of Stage 1 randomization to a treatment arm
Period: Overall Study
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures | Not Randomized to Treatment
Started | 149 | 288 | 265 | 282 | 242 | 13 | 509
Completed | 0 | 140 | 134 | 131 (96 of these completed at least 1 coaching check-in addition to completing 5 sessions of CBM-I) | 154 | 0 | 0
Not Completed | 149 | 148 | 131 | 151 | 88 | 13 | 509

BASELINE CHARACTERISTICS:
Population: A few participants were excluded from analyses during data cleaning due to concerns about integrity of their data, hence the # of baseline participants is slightly below the enrollment #.
  Participants not randomized to treatment often did not complete demographic information and were not included in analyses.
Groups:
- Received CBM-I and Not Classified as High/Low Risk for Attrition: This group started treatment (and had been randomized to CBM-I) but did not complete Session 1 of CBM-I training plus assessments, so was not classified as high/low risk for attrition and thus not randomized for Stage 2 of SMART design
- Removed From Analyses: 5 participants were removed from analyses as there were concerns with the integrity of their data
- Total: Total of all reporting groups
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures | Not Randomized to Treatment | Removed From Analyses | Total
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13 | 0 | 5 | 1239
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.16 (12.09) | 37.2 (12.33) | 34.24 (11.13) | 34.37 (11.9) | 35.09 (12.3) | 31.54 (10.44) |  | 28.50 (3.32) | 35.09 (11.97)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 112 | 237 | 217 | 231 | 194 | 11 |  | 1 | 1003
  Male | 33 | 45 | 38 | 43 | 41 | 2 |  | 3 | 205
  Transgender | 0 | 0 | 2 | 2 | 1 | 0 |  | 0 | 5
  Transgender Female | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0
  Transgender Male | 0 | 1 | 2 | 0 | 1 | 0 |  | 0 | 4
  Other | 2 | 4 | 4 | 4 | 2 | 0 |  | 0 | 16
  Prefer not to answer | 1 | 1 | 0 | 1 | 2 | 0 |  | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 22 | 40 | 31 | 38 | 30 | 3 |  | 0 | 164
  Ethnicity: Not Hispanic or Latino | 118 | 230 | 224 | 236 | 201 | 10 |  | 2 | 1021
  Ethnicity: Unknown | 3 | 7 | 4 | 5 | 2 | 0 |  | 1 | 22
  Ethnicity: Prefer not to answer | 5 | 11 | 4 | 2 | 8 | 0 |  | 2 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian/Alaska Native | 1 | 3 | 3 | 1 | 1 | 0 |  | 0 | 9
  Race: Black/African origin | 12 | 31 | 27 | 19 | 31 | 2 |  | 0 | 122
  Race: East Asian | 4 | 5 | 7 | 11 | 9 | 0 |  | 1 | 37
  Race: Native Hawaiian/Pacific Islander | 1 | 2 | 1 | 0 | 0 | 0 |  | 0 | 4
  Race: South Asian | 3 | 4 | 6 | 5 | 7 | 2 |  | 2 | 29
  Race: White/European origin | 95 | 211 | 185 | 212 | 179 | 8 |  | 1 | 891
  Race: More than one race | 18 | 18 | 22 | 24 | 5 | 0 |  | 0 | 87
  Race: Other or Unknown | 12 | 10 | 10 | 6 | 4 | 1 |  | 0 | 43
  Race: Prefer not to answer | 2 | 4 | 2 | 3 | 5 | 0 |  | 1 | 17
Country [Count of Participants; unit: Participants] — Countries with fewer than 10 participants in the Stage 1 randomized sample (n = 1,614) were collapsed into Other.
  Participants
    United States | 133 | 256 | 251 | 259 | 214 | 12 |  | 2 | 1127
    Australia | 4 | 17 | 8 | 10 | 12 | 1 |  | 0 | 52
    United Kingdom | 3 | 4 | 1 | 0 | 4 | 0 |  | 1 | 13
    Canada | 3 | 4 | 1 | 1 | 3 | 0 |  | 0 | 12
    Other | 4 | 7 | 2 | 11 | 7 | 0 |  | 1 | 32
    Prefer not to answer | 1 | 0 | 0 | 0 | 1 | 0 |  | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Recognition Ratings (Positive Interpretation Bias)
Description: To measure interpretation bias, participants will read ambiguous scenarios with titles, after which they will see the titles of each scenario, followed by 4 interpretations of the scenario: 1 positive and threat related, 1 negative and threat related, 1 positive and threat unrelated, and 1 negative and threat unrelated. Participants will rate each interpretation based on how similar in meaning it is to the original scenario on a 4-point scale ranging from 1 to 4. The mean of the positive, threat-related ratings index positive interpretation bias. Higher scores represent a more positive interpretation bias.
Time Frame: Baseline, and after session 3 (2-3 weeks following baseline), session 5 (~2 weeks after session 3), & at 2-month follow-up (~ 2 months after session 5). Measure will be completed immediately following that day's training session.
Population: A few participants were excluded from analyses during data cleaning due to concerns about integrity of their data, hence the # of analyzed participants is slightly below the enrollment #.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment: number analyzed (Participants) | 148 | 287 | 263 | 281 | 240 | 13
  Baseline assessment | 2.40 (0.47) | 2.29 (0.53) | 2.29 (0.54) | 2.30 (0.53) | 2.33 (0.54) | 2.40 (0.60)
  Session 3 assessment: number analyzed (Participants) | 0 | 179 | 172 | 158 | 178 | 0
  Session 3 assessment |  | 2.89 (0.44) | 2.84 (0.48) | 2.92 (0.49) | 2.39 (0.57) |
  Session 5 assessment: number analyzed (Participants) | 0 | 138 | 132 | 129 | 153 | 0
  Session 5 assessment |  | 2.83 (0.52) | 2.92 (0.44) | 2.86 (0.50) | 2.42 (0.55) |
  Follow-up assessment: number analyzed (Participants) | 0 | 128 | 113 | 109 | 130 | 0
  Follow-up assessment |  | 2.71 (0.47) | 2.80 (0.46) | 2.75 (0.54) | 2.48 (0.53) |
Statistical Analysis 1: Comparison: Received CBM-I and Not Classified as High/Low Risk for Attrition vs Received CBM-I and Classified Low Attrition vs Received CBM-I and Classified High Attrition and no Coach Given vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; Intent-to-treat (ITT) analysis of Stage 1 randomization to CBM-I vs. psychoeducation. To correct for sampling bias (i.e., "CBM-I, high attrition, coach" received coaching, whereas psychoeducation did not receive coaching), "CBM-I, high attrition, coach" participants were excluded and replaced with an equal number of "CBM-I, high attrition, no coach" participants (using bootstrap resampling). The corrected ITT analysis sample included 1,234 participants (980 in CBM-I, 254 in psychoeducation); Test type: Superiority; Mixed Models Analysis; We compared the two groups in a piecewise linear multilevel model (one slope during treatment, one during follow-up), controlling for income and age; Mean Difference (Net) = 1.10, 95% CI 2-sided [1.04 to 1.16], Standard Deviation 0.03 — From the model (run in Bayesian with non-informative priors), we report the between-group SMD (with empirical SD & 95% bootstrap confidence interval) at Session 5 (at mean income & age), adjusted for baseline differences & using pooled baseline SD
Statistical Analysis 2: Comparison: Received CBM-I and Classified High Attrition and no Coach Given vs Received CBM-I and Classified High Attrition and Given a Coach; Analysis of Stage 2 randomization of CBM-I participants classified as high risk for attrition to supplemental coaching vs. no coaching. The analysis sample included 544 participants (263 in "CBM-I, high attrition, no coach"; 281 in "CBM-I, high attrition, coach"); Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.43 to 0.20], Standard Deviation 0.16 — From the model (run in Bayesian with non-informative priors), we report the between-group SMD (with empirical SD & 95% HPD credible interval) at Session 5 (at mean income & age), adjusted for baseline differences & using pooled baseline SD

2. Primary Outcome: Change in Recognition Ratings (Negative Interpretation Bias)
Description: To measure interpretation bias, participants will read ambiguous scenarios with titles, after which they will see the titles of each scenario, followed by 4 interpretations of the scenario: 1 positive and threat related, 1 negative and threat related, 1 positive and threat unrelated, and 1 negative and threat unrelated. Participants will rate each interpretation based on how similar in meaning it is to the original scenario on a 4-point scale ranging from 1 to 4. The mean of the negative, threat-related ratings index negative interpretation bias. Higher scores represent a more negative interpretation bias.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CBM-I, Not Classified as High/Low Risk for Attrition: This group started treatment (and had been randomized to CBM-I) but did not complete Session 1 of CBM-I training plus assessments, so was not classified as high/low risk for attrition and thus not randomized for Stage 2 of SMART design
Arm/Group | CBM-I, Not Classified as High/Low Risk for Attrition | CBM-I, Low Attrition | CBM-I, High Attrition, no Coach | CBM-I, High Attrition, Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment: number analyzed (Participants) | 148 | 287 | 263 | 281 | 240 | 13
  Baseline assessment | 2.78 (0.53) | 2.90 (0.54) | 2.96 (0.51) | 2.94 (0.55) | 2.89 (0.50) | 2.70 (0.60)
  Session 3 assessment: number analyzed (Participants) | 0 | 180 | 172 | 158 | 178 | 0
  Session 3 assessment |  | 2.56 (0.56) | 2.49 (0.55) | 2.46 (0.58) | 2.87 (0.55) |
  Session 5 assessment: number analyzed (Participants) | 0 | 138 | 132 | 129 | 153 | 0
  Session 5 assessment |  | 2.58 (0.55) | 2.53 (0.56) | 2.56 (0.52) | 2.74 (0.59) |
  Follow-up assessment: number analyzed (Participants) | 0 | 128 | 113 | 109 | 130 | 0
  Follow-up assessment |  | 2.55 (0.55) | 2.48 (0.56) | 2.43 (0.58) | 2.68 (0.58) |
Statistical Analysis 1: Comparison: CBM-I, Not Classified as High/Low Risk for Attrition vs CBM-I, Low Attrition vs CBM-I, High Attrition, no Coach vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.63, 95% CI 2-sided [-0.69 to -0.57], Standard Deviation 0.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CBM-I, High Attrition, no Coach vs CBM-I, High Attrition, Coach; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.26 to 0.39], Standard Deviation 0.17 — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Change in Brief Bodily Sensations Interpretations Questionnaire (Benign Interpretation Bias)
Description: To assess interpretation change, participants are presented with ambiguous events and then asked to rate three alternative explanations for why the event might have occurred on a 5-point scale ranging from 0 to 4. One option is always negative and threat related, whereas the other options are mixed in valence but threat unrelated. We computed the mean of the threat-unrelated ratings as an index of benign interpretation bias. Higher scores represent a more benign interpretation bias.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBM-I, Not Classified as High/Low Risk for Attrition | CBM-I, Low Attrition | CBM-I, High Attrition, no Coach | CBM-I, High Attrition, Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment | 2.04 (0.55) | 2.00 (0.53) | 2.13 (0.49) | 2.05 (0.52) | 2.07 (0.55) | 2.23 (0.38)
  Session 3 assessment: number analyzed (Participants) | 0 | 177 | 171 | 157 | 177 | 0
  Session 3 assessment |  | 2.25 (0.55) | 2.38 (0.53) | 2.36 (0.52) | 2.20 (0.51) |
  Session 5 assessment: number analyzed (Participants) | 0 | 138 | 132 | 129 | 153 | 0
  Session 5 assessment |  | 2.34 (0.62) | 2.51 (0.52) | 2.45 (0.53) | 2.19 (0.58) |
  Follow-up assessment: number analyzed (Participants) | 0 | 128 | 112 | 109 | 130 | 0
  Follow-up assessment |  | 2.31 (0.56) | 2.35 (0.58) | 2.36 (0.55) | 2.23 (0.61) |
Statistical Analysis 1: Comparison: CBM-I, Not Classified as High/Low Risk for Attrition vs CBM-I, Low Attrition vs CBM-I, High Attrition, no Coach vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.48, 95% CI 2-sided [0.42 to 0.54], Standard Deviation 0.03; From the model (run in Bayesian with non-informative priors), we report the between-group SMD (with empirical SD & 95% bootstrap confidence interval) at Session 5 (at mean income & age), adjusted for baseline differences & using pooled baseline SD
Statistical Analysis 2: Comparison: CBM-I, High Attrition, no Coach vs CBM-I, High Attrition, Coach; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.23 to 0.39], Standard Deviation 0.16 — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Change in Brief Bodily Sensations Interpretations Questionnaire (Negative Interpretation Bias)
Description: To assess interpretation change, participants are presented with ambiguous events and then asked to rate three alternative explanations for why the event might have occurred on a 5-point scale ranging from 0 to 4. One option is always negative and threat related, whereas the other options are mixed in valence but threat unrelated. We computed the mean of the negative, threat-related ratings as an index of negative interpretation bias. Higher scores represent a more negative interpretation bias.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBM-I, Not Classified as High/Low Risk for Attrition | CBM-I, Low Attrition | CBM-I, High Attrition, no Coach | CBM-I, High Attrition, Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment | 1.42 (0.83) | 1.61 (0.86) | 1.52 (0.81) | 1.58 (0.82) | 1.61 (0.81) | 1.35 (0.94)
  Session 3 assessment: number analyzed (Participants) | 0 | 176 | 171 | 157 | 177 | 0
  Session 3 assessment |  | 0.93 (0.80) | 0.85 (0.66) | 0.85 (0.71) | 1.36 (0.81) |
  Session 5 assessment: number analyzed (Participants) | 0 | 138 | 132 | 129 | 153 | 0
  Session 5 assessment |  | 0.81 (0.68) | 0.77 (0.68) | 0.83 (0.70) | 1.24 (0.78) |
  Follow-up assessment: number analyzed (Participants) | 0 | 128 | 112 | 109 | 130 | 0
  Follow-up assessment |  | 0.78 (0.62) | 0.79 (0.62) | 0.69 (0.57) | 1.16 (0.77) |
Statistical Analysis 1: Comparison: CBM-I, Not Classified as High/Low Risk for Attrition vs CBM-I, Low Attrition vs CBM-I, High Attrition, no Coach vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.55, 95% CI 2-sided [-0.60 to -0.51], Standard Deviation 0.02 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CBM-I, High Attrition, no Coach vs CBM-I, High Attrition, Coach; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.23 to 0.27], Standard Deviation 0.13 — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Change in Overall Anxiety Severity and Impairment Scale
Description: This 5-item measure of anxiety symptom severity and impairment has good psychometric properties, shows treatment sensitivity, and is valid in community and clinical samples. Item range = 0 to 4 (5-point scale). Total scale range = 0-20, with a higher score indicating more severe anxiety. Average item scores are reported below.
Time Frame: Baseline, and after sessions 1,2, 3, 4, 5 (sessions will be spaced ~1 week apart) & at 2-month follow-up (~2 months after session 5). Session 1 occurs ~0-7 days after baseline. Measure will be completed immediately following that day's training session.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBM-I, Not Classified as High/Low Risk for Attrition | CBM-I, Low Attrition | CBM-I, High Attrition, no Coach | CBM-I, High Attrition, Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment | 2.28 (0.75) | 2.32 (0.71) | 2.31 (0.67) | 2.34 (0.67) | 2.31 (0.68) | 2.62 (0.79)
  Session 1 assessment: number analyzed (Participants) | 1 | 287 | 263 | 281 | 240 | 0
  Session 1 assessment | 2.00 (NA) — 1 Participant | 2.22 (0.73) | 2.15 (0.75) | 2.21 (0.72) | 2.24 (0.73) |
  Session 2 assessment: number analyzed (Participants) | 0 | 207 | 192 | 187 | 187 | 0
  Session 2 assessment |  | 1.75 (0.74) | 1.71 (0.74) | 1.79 (0.75) | 1.92 (0.75) |
  Session 3 assessment: number analyzed (Participants) | 0 | 185 | 173 | 161 | 181 | 0
  Session 3 assessment |  | 1.80 (0.80) | 1.72 (0.79) | 1.84 (0.74) | 2.00 (0.78) |
  Session 4 assessment: number analyzed (Participants) | 0 | 150 | 145 | 142 | 161 | 0
  Session 4 assessment |  | 1.63 (0.84) | 1.48 (0.80) | 1.53 (0.78) | 1.85 (0.90) |
  Session 5 assessment: number analyzed (Participants) | 0 | 140 | 132 | 131 | 153 | 0
  Session 5 assessment |  | 1.58 (0.78) | 1.50 (0.78) | 1.62 (0.80) | 1.77 (0.85) |
  Follow-up assessment: number analyzed (Participants) | 0 | 129 | 115 | 110 | 130 | 0
  Follow-up assessment |  | 1.59 (0.79) | 1.56 (0.87) | 1.60 (0.79) | 1.68 (0.81) |
Statistical Analysis 1: Comparison: CBM-I, Not Classified as High/Low Risk for Attrition vs CBM-I, Low Attrition vs CBM-I, High Attrition, no Coach vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.41, 95% CI 2-sided [-0.46 to -0.37], Standard Deviation 0.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CBM-I, High Attrition, no Coach vs CBM-I, High Attrition, Coach; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.23 to 0.32], Standard Deviation 0.14 — [estimate comment as in outcome 1, analysis 2]

6. Primary Outcome: Change in Depression, Anxiety, Stress Scales-Short Form: Anxiety Subscale
Description: This 7-item measure of anxiety symptoms has good psychometric properties, shows treatment sensitivity, and is valid in community and clinical samples. Item range = 0 to 3 (4-point scale). Total DASS-21 anxiety subscale range = 0-21 (multiplied by 2 for DASS-42 = 0-42), with a higher score indicating more severe anxiety symptoms. Average item scores are reported below.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBM-I, Not Classified as High/Low Risk for Attrition | CBM-I, Low Attrition | CBM-I, High Attrition, no Coach | CBM-I, High Attrition, Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
units on a scale
  Baseline assessment | 1.61 (0.55) | 1.58 (0.53) | 1.65 (0.54) | 1.65 (0.53) | 1.65 (0.52) | 1.71 (0.64)
  Session 3 assessment: number analyzed (Participants) | 0 | 185 | 172 | 161 | 181 | 0
  Session 3 assessment |  | 1.01 (0.61) | 0.98 (0.62) | 1.07 (0.62) | 1.19 (0.64) |
  Session 5 assessment: number analyzed (Participants) | 0 | 140 | 132 | 131 | 153 | 0
  Session 5 assessment |  | 0.89 (0.58) | 0.83 (0.57) | 0.89 (0.62) | 1.03 (0.67) |
  Follow-up assessment: number analyzed (Participants) | 0 | 129 | 115 | 109 | 130 | 0
  Follow-up assessment |  | 0.82 (0.57) | 0.80 (0.63) | 0.80 (0.64) | 0.97 (0.62) |
Statistical Analysis 1: Comparison: CBM-I, Not Classified as High/Low Risk for Attrition vs CBM-I, Low Attrition vs CBM-I, High Attrition, no Coach vs Psychoeducation vs Psychoeducation, Lacking Classification Measures; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.39 to -0.27], Standard Deviation 0.03 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CBM-I, High Attrition, no Coach vs CBM-I, High Attrition, Coach; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.14 to 0.48], Standard Deviation 0.16 — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change in Depression Comorbid Symptoms
Description: The Patient Health Questionnaire 2 (PHQ-2) inquires about the frequency of depressed mood and anhedonia. A score of 3 or higher on the Patient Health Questionnaire-2 (PHQ-2) is considered an indication of major depressive disorder. The PHQ-2 is a two-question screening tool that asks how often a person has experienced depressed mood or anhedonia over the past two weeks. The score range is 0-6, with higher scores indicating more frequent symptoms, and response options 0-3 for each question where 0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day.
Time Frame: as for outcome 1
Population: Some weeks have less participants reported than overall number analyzed because of attrition - participants did not fill out the survey and thus we do not have data to report on all participants across all weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 286 | 263 | 281 | 241 | 13
  Baseline | 2.77 (0.86) | 2.76 (0.90) | 2.68 (0.93) | 2.77 (0.91) | 2.78 (0.89) | 2.92 (0.95)
  Session 3: number analyzed (Participants) | 0 | 177 | 171 | 158 | 178 | 0
  Session 3 |  | 2.35 (0.92) | 2.22 (0.86) | 2.32 (0.90) | 2.49 (0.96) |
  Session 5: number analyzed (Participants) | 0 | 140 | 132 | 130 | 153 | 0
  Session 5 |  | 2.15 (0.92) | 2.12 (0.90) | 2.13 (0.90) | 2.36 (0.97) |
  2-month Follow-up: number analyzed (Participants) | 0 | 129 | 112 | 109 | 130 | 0
  2-month Follow-up |  | 2.15 (0.91) | 2.00 (0.93) | 2.00 (0.89) | 2.09 (0.88) |

8. Secondary Outcome: Change in Alcohol Use Comorbid Symptoms
Description: The Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) is a 3-item alcohol screen that can help identify persons who are hazardous drinkers or have active alcohol use disorders. The AUDIT has 10 questions and the possible responses to each question are scored 0, 1, 2, 3 or 4, with the exception of questions 9 and 10 which have possible responses of 0, 2 and 4. The range of possible scores is from 0 to 40 where 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 288 | 263 | 280 | 240 | 13
  Baseline | 0.92 (0.82) | 0.90 (0.84) | 0.94 (0.86) | 0.95 (0.79) | 0.90 (0.89) | 0.64 (0.73)
  Session 3: number analyzed (Participants) | 0 | 177 | 171 | 158 | 178 | 0
  Session 3 |  | 0.88 (0.89) | 0.92 (0.83) | 0.80 (0.73) | 0.84 (0.85) |
  Session 5: number analyzed (Participants) | 0 | 140 | 132 | 130 | 153 | 0
  Session 5 |  | 0.75 (0.75) | 0.85 (0.77) | 0.71 (0.73) | 0.78 (0.80) |
  2-month Follow-up: number analyzed (Participants) | 0 | 129 | 112 | 109 | 129 | 0
  2-month Follow-up |  | 0.78 (0.80) | 0.80 (0.70) | 0.59 (0.62) | 0.71 (0.80) |

9. Secondary Outcome: Change in Wellness Measures - Optimism
Description: Items 3 and 7 from the Life Orientation Test-Revised (LOT-R) assess generalized optimism versus pessimism.
  Responses include: 0 = Strongly disagree, 1 = Disagree, 2 = Neutral, 3 = Agree, and 4 = Strongly agree, plus Prefer not to answer. Total aggregate scores range from 0 to 4 by taking the mean of the 2 items.
  Higher scores indicate lower optimism/higher pessimism. We calculate participants' optimism scores by taking the mean of the two items, and we are reporting these mean optimism scores below.
  Questions are:
  If something can go wrong with me, it will. I hardly ever expect things to go my way.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 286 | 263 | 281 | 241 | 13
  Baseline | 1.33 (1.00) | 1.40 (0.97) | 1.39 (0.96) | 1.45 (1.02) | 1.29 (0.97) | 1.85 (1.43)
  Session 3: number analyzed (Participants) | 0 | 175 | 171 | 157 | 178 | 0
  Session 3 |  | 1.82 (0.94) | 1.82 (1.05) | 1.79 (1.07) | 1.52 (0.98) |
  Session 5: number analyzed (Participants) | 0 | 139 | 132 | 129 | 152 | 0
  Session 5 |  | 1.85 (1.03) | 1.97 (1.06) | 1.82 (1.01) | 1.57 (0.97) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 129 | 0
  2-month Follow-up |  | 1.93 (1.03) | 1.84 (1.08) | 1.95 (1.07) | 1.65 (0.93) |

10. Secondary Outcome: Change in Wellness Measures - Growth Mindset
Description: Items 1, 5, and 7 from the Growth Mindset Measure were administered to measure changes in thinking styles (altered from the original items that reference intelligence).
  Responses include: 0 = Strongly disagree, 1 = Disagree, 2 = Neutral, 3 = Agree, and 4 = Strongly agree, plus Prefer not to answer. Total aggregate scores can range from 0 to 4 by taking the mean of the 3 items.
  Higher scores indicate a lack of a growth mindset (AKA more negative outcome). We calculate participants' growth mindset scores by taking the mean of the two items, and we are reporting these mean growth mindset scores below.
  Questions are:
  You can learn new things, but you can't really change how you think. No matter how much you have been thinking a particular way, you can always change it quite a bit.
  You can always substantially change how you think.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 241 | 13
  Baseline | 2.17 (0.57) | 2.14 (0.50) | 2.12 (0.55) | 2.10 (0.51) | 2.13 (0.53) | 2.13 (0.44)
  Session 3: number analyzed (Participants) | 0 | 177 | 171 | 157 | 178 | 0
  Session 3 |  | 2.29 (0.53) | 2.33 (0.53) | 2.27 (0.47) | 2.20 (0.49) |
  Session 5: number analyzed (Participants) | 0 | 139 | 132 | 129 | 152 | 0
  Session 5 |  | 2.29 (0.53) | 2.34 (0.51) | 2.25 (0.53) | 2.28 (0.52) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 129 | 0
  2-month Follow-up |  | 2.22 (0.47) | 2.25 (0.52) | 2.26 (0.46) | 2.25 (0.50) |

11. Secondary Outcome: Change in Wellness Measures - Self-efficacy
Description: Items 2, 6, and 7 from the New General Self-Efficacy Scale (NGSES) will be administered to measure self-efficacy. Item range = 0 to 4. Total aggregate scores can range from 0 to 4 by taking the mean of the 3 items.
  Higher scores indicate more self-efficacy. We calculate participants' self-efficacy scores by taking the mean of the 3 items.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 241 | 13
  Baseline | 2.27 (0.93) | 2.27 (0.92) | 2.37 (0.83) | 2.22 (0.93) | 2.20 (0.93) | 2.15 (1.04)
  Session 3: number analyzed (Participants) | 0 | 177 | 171 | 157 | 178 | 0
  Session 3 |  | 2.71 (0.84) | 2.75 (0.85) | 2.59 (0.81) | 2.41 (0.83) |
  Session 5: number analyzed (Participants) | 0 | 139 | 132 | 129 | 152 | 0
  Session 5 |  | 2.77 (0.81) | 2.75 (0.79) | 2.74 (0.84) | 2.57 (0.88) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 129 | 0
  2-month Follow-up |  | 2.75 (0.75) | 2.82 (0.74) | 2.75 (0.78) | 2.58 (0.80) |

12. Secondary Outcome: Change in Wellness Measures - Life Satisfaction
Description: Single-Item Life Satisfaction measure will be administered to measure overall satisfaction with one's life.
  Participants are asked "All things considered, how satisfied are you with your life as a whole?" and can choose from the following options, with lower scores being more dissatisfied with life (AKA more negative):
  0 (Completely dissatisfied)
  1 2 3 4 5 6 7 8 9 10 (Completely satisfied) Prefer not to answer
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 262 | 280 | 241 | 13
  Baseline | 4.71 (2.28) | 4.77 (2.22) | 5.09 (2.16) | 4.95 (2.14) | 5.01 (2.18) | 4.31 (2.50)
  Session 3: number analyzed (Participants) | 0 | 177 | 171 | 158 | 178 | 0
  Session 3 |  | 5.69 (2.21) | 5.75 (2.05) | 5.94 (1.99) | 5.28 (2.13) |
  Session 5: number analyzed (Participants) | 0 | 140 | 132 | 129 | 152 | 0
  Session 5 |  | 5.81 (2.32) | 6.00 (2.08) | 6.01 (1.91) | 5.79 (2.05) |
  2-month Follow-up: number analyzed (Participants) | 0 | 129 | 112 | 110 | 130 | 0
  2-month Follow-up |  | 5.71 (2.16) | 6.12 (2.05) | 6.14 (2.03) | 5.76 (1.91) |

13. Secondary Outcome: Change in Mechanisms Underlying Bias Change - Cognitive Flexibility
Description: Item 14 of the Cognitive Flexibility Inventory (CFI) will be administered to measure cognitive flexibility.
  Participants are asked "I often look at a situation from different viewpoints." with response options as follows, with higher scores indicating more cognitive flexibility (AKA more positive outcome):
  1. = Strongly disagree
  2. = Disagree
  3. = Somewhat disagree
  4. = Neutral
  5. = Somewhat agree
  6. = Agree
  7. = Strongly agree Prefer not to answer
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 240 | 13
  Baseline | 5.20 (1.41) | 5.20 (1.43) | 5.25 (1.38) | 5.17 (1.51) | 5.04 (1.44) | 5.54 (1.05)
  Session 3: number analyzed (Participants) | 0 | 175 | 171 | 157 | 177 | 0
  Session 3 |  | 5.41 (1.31) | 5.60 (1.33) | 5.41 (1.35) | 5.36 (1.24) |
  Session 5: number analyzed (Participants) | 0 | 139 | 132 | 129 | 150 | 0
  Session 5 |  | 5.40 (1.40) | 5.61 (1.35) | 5.52 (1.23) | 5.33 (1.26) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 130 | 0
  2-month Follow-up |  | 5.59 (1.15) | 5.57 (1.19) | 5.57 (1.20) | 5.47 (1.26) |

14. Secondary Outcome: Change in Mechanisms Underlying Bias Change - Experiential Avoidance
Description: Item 11 from the Comprehensive Assessment of ACT processes (CompACT) will be administered to measure experiential avoidance.
  Participants are asked "I am willing to fully experience whatever thoughts, feelings, and sensations come up for me, without trying to change them." with response options as follows, with higher scores indicating less avoidance (AKA more positive outcome):
  1. = Strongly disagree
  2. = Disagree
  3. = Somewhat disagree
  4. = Neutral
  5. = Somewhat agree
  6. = Agree
  7. = Strongly agree Prefer not to answer
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 241 | 13
  Baseline | 4.05 (1.75) | 3.78 (1.66) | 3.89 (1.63) | 3.85 (1.64) | 3.80 (1.55) | 3.85 (1.41)
  Session 3: number analyzed (Participants) | 0 | 175 | 171 | 156 | 176 | 0
  Session 3 |  | 4.33 (1.60) | 4.44 (1.60) | 3.94 (1.57) | 4.14 (1.53) |
  Session 5: number analyzed (Participants) | 0 | 138 | 132 | 129 | 150 | 0
  Session 5 |  | 4.56 (1.55) | 4.72 (1.41) | 4.43 (1.56) | 4.25 (1.48) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 130 | 0
  2-month Follow-up |  | 4.58 (1.51) | 4.73 (1.54) | 4.17 (1.61) | 4.35 (1.43) |

15. Secondary Outcome: Change in Mechanisms Underlying Bias Change - Cognitive Reappraisal
Description: Items 7 and 10 from the Emotion Regulation Questionnaire (ERQ) will be administered to measure cognitive reappraisal.
  Participants are given two statements - "When I want to feel more positive emotion, I change the way I'm thinking about the situation" and "When I want to feel less negative emotion, I change the way I'm thinking about the situation" - with response options as follows, with higher scores indicating more reappraisal (AKA more positive outcome):
  1. = Strongly disagree
  2. = Disagree
  3. = Somewhat disagree
  4. = Neutral
  5. = Somewhat agree
  6. = Agree
  7. = Strongly agree Prefer not to answer
  Total aggregate scores can range from 0 to 7 by taking the mean of the two items. We calculate participants' Cognitive reappraisal scores by taking the mean of the two items, and we are reporting these mean Cognitive reappraisal scores below.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 241 | 13
  Baseline | 4.41 (1.57) | 4.28 (1.49) | 4.34 (1.42) | 4.29 (1.41) | 4.14 (1.36) | 4.65 (1.05)
  Session 3: number analyzed (Participants) | 0 | 175 | 171 | 157 | 177 | 0
  Session 3 |  | 4.90 (1.25) | 4.81 (1.44) | 4.79 (1.28) | 4.59 (1.33) |
  Session 5: number analyzed (Participants) | 0 | 138 | 132 | 129 | 151 | 0
  Session 5 |  | 5.11 (1.28) | 4.95 (1.20) | 4.89 (1.32) | 4.87 (1.29) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 130 | 0
  2-month Follow-up |  | 5.00 (1.20) | 4.96 (1.18) | 5.01 (1.18) | 4.92 (1.11) |

16. Secondary Outcome: Change in Mechanisms Underlying Bias Change - Intolerance of Uncertainty
Description: Items 1 and 7 from the Intolerance of Uncertainty Scale-Short Form (IUS-12) will be administered to measure intolerance of uncertainty. Item range = 1 to 7. Total range for aggregated 2 items = 2-14, with a higher score indicating more intolerance of uncertainty.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 287 | 263 | 281 | 241 | 13
  Baseline | 5.42 (1.27) | 5.57 (1.11) | 5.56 (1.14) | 5.65 (1.12) | 5.53 (1.23) | 5.62 (1.16)
  Session 3: number analyzed (Participants) | 0 | 175 | 171 | 157 | 177 | 0
  Session 3 |  | 5.22 (1.20) | 5.18 (1.19) | 5.29 (1.17) | 5.44 (1.20) |
  Session 5: number analyzed (Participants) | 0 | 137 | 132 | 129 | 151 | 0
  Session 5 |  | 5.00 (1.37) | 5.08 (1.14) | 5.03 (1.21) | 5.25 (1.22) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 112 | 109 | 129 | 0
  2-month Follow-up |  | 5.10 (1.31) | 5.16 (1.20) | 5.02 (1.20) | 5.26 (1.19) |

17. Secondary Outcome: Change in Anxiety and Identity Circles
Description: We will assess change in the extent anxiety is viewed as central to the person's self-concept.
  Participants are asked "To what extent is your anxiety a central part of who you are currently?" and provided with 5 images of two circles, one labeled "My Anxiety" and one labeled "Me", where the circles start off not touching at all and get increasingly closer/overlapped, with the last image having the circles fully overlapped. We code these 5 images as 0 = No overlap, 1 = overlapped about 25%, 2 = overlapped about 50%, 3 = overlapped about 75%, 4 = Fully overlapped; higher scores indicate that anxiety is more central to the person's self-concept, and lower scores indicate that the person does not identify themself with their anxiety.
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures
Number analyzed (Participants) | 148 | 288 | 263 | 281 | 241 | 13
score on a scale
  Baseline: number analyzed (Participants) | 148 | 288 | 263 | 280 | 241 | 12
  Baseline | 2.48 (0.93) | 2.55 (0.90) | 2.51 (0.88) | 2.56 (0.85) | 2.49 (0.98) | 2.42 (0.79)
  Session 3: number analyzed (Participants) | 0 | 184 | 173 | 161 | 181 | 0
  Session 3 |  | 1.93 (0.93) | 1.86 (0.92) | 2.01 (0.90) | 2.12 (0.95) |
  Session 5: number analyzed (Participants) | 0 | 139 | 132 | 131 | 153 | 0
  Session 5 |  | 1.61 (1.00) | 1.69 (0.79) | 1.75 (0.99) | 1.83 (0.94) |
  2-month Follow-up: number analyzed (Participants) | 0 | 128 | 115 | 110 | 130 | 0
  2-month Follow-up |  | 1.57 (0.88) | 1.54 (0.85) | 1.57 (0.89) | 1.78 (1.01) |

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored throughout the study, through study completion (during the 5-6 weeks of active study sessions and at 2 month follow-up).
Description: No difference
Groups:
- Psychoeducation: Online psychoeducation about anxiety Online psychoeducation about anxiety: Participants will review webpages that describe information about symptoms and causes of anxiety, including the nature of biased thinking in anxiety
Arm/Group | Received CBM-I and Not Classified as High/Low Risk for Attrition | Received CBM-I and Classified Low Attrition | Received CBM-I and Classified High Attrition and no Coach Given | Received CBM-I and Classified High Attrition and Given a Coach | Psychoeducation | Psychoeducation, Lacking Classification Measures | Not Randomized to Treatment
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/288 | 0/265 | 0/282 | 0/242 | 0/13 | 0/509
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/288 | 0/265 | 0/282 | 0/242 | 0/13 | 0/509
Other Adverse Events (participants affected / at risk) | 0/149 | 0/288 | 0/265 | 0/282 | 0/242 | 0/13 | 0/509

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT03498651/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03498651/ICF_001.pdf